CLINICAL TRIAL: NCT06950138
Title: Efficacy of Triticum Aestivum Over Vascular Function in Mexican Obese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2023-130-177
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Vascular Risk
Keywords: Triticum aestivum; Obesity; Arterial stiffness; Flow-mediated dilatation; Wave pulse velocity
MeSH Terms: conditions — Obesity | interventions — Flour; Magnesium Oxide

STUDY DESIGN:
Intervention Model Description: Intervention group that received 1 capsule of 500 mg of Triticum aestivum every 12 hours for 120 days (n=10), and a control group that received placebo with the same organoleptic characteristics for the same period (n=10). Both groups received general lifestyle and dietary recommendations.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Stratified random sampling with a closed envelope, random number assigned by software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triticum aestivum (Active Comparator): A group of 20 patients with a diagnosis of obesity without current treatment or other associated pathologies, who will receive 500 mg of triticum aestivum orally every 12 hours for 120 days.
- Calcined magnesia (Placebo Comparator): A group of 20 patients with a diagnosis of obesity without current treatment or other associated pathologies, who will recive 500 mg of calcined magnesia oraly every 12 hours for 120 days.
  Interventions: Drug: calcined magnesia

INTERVENTIONS:
Drug: Triticum aestivum — During the intervention period, the aim is to evaluate changes in the patient's vascular function.
Drug: calcined magnesia — During the intervention period, the aim is to evaluate changes in the patient's vascular function.
  Other Names: Magnesium oxide
  Arms: Calcined magnesia

SUMMARY:
This study aims to evaluate the efficacy of Triticum aestivum as a treatment for improving the vascular function in Mexican obese patients. We conducted a triple-blind, randomized, placebo controlled clinical trial, involving obese individuals from the metropolitan area of Guadalajara. The participants were randomly assigned to either Triticum aestivum (intervention group) or placebo supplementation (control). The primary outcome measures were those related with the vascular function using non-invasive methods such as flow-mediated dilation and wave pulse velocity measurements. Secondary outcomes included changes in anthropometric or clinical measures, laboratory results and molecular markers (endothelin-1 and nitric oxide). Data were collected at baseline and after the intervention period. Statistical analyses were performed to determine the significance of the observed changes.

DETAILED DESCRIPTION:
Background:

Obesity is a multifactorial disease highly prevalent among Mexican population. It is closely related to the maintenance of a pro-inflammatory syndrome. This promotes the development of physiopathological mechanisms that support and perpetuate the vascular disfunction which can contribute to the development of cardiovascular disease.

The vascular disfunction is closely related to the impaired endothelial function and increase arterial stiffness. Currently there is no specific treatment for vascular disfunction. Triticum aestivum, or wheatgrass, is a known plant, used primary for its anti-inflammatory and antioxidant properties. This trial aim to investigate the potential health benefits in vascular function of Mexican obese patients. Triticum aestivum is rich in fibers, vitamins, minerals, and polyphenols. Polyphenols, such as flavonoids have antioxidant and anti-inflammatory properties. The flavonoids in wheat grass can scavenge free radicals, preventing cellular damage and preserving endothelial function. In addition, flavonoids have demonstrated anti-inflammatory effects, modulating inflammatory processes within the vascular system. Moreover, the flavonoids can contribute to a improve lipid profile by reducing low density cholesterol levels.

Objetive:

Evaluate the efficacy of Triticum aestivum versus placebo over the vascular function of Mexican obese patients.

Study Design:

A randomized, triple-blind, placebo-controlled clinical trial in Mexican patients with obesity from the metropolitan area of Guadalajara diagnosed according to WHO criteria, who agreed to participate in the protocol through informed consent, randomly assigned to two groups: an intervention group that will receive 1 capsule of 500 mg of Triticum aestivum every 12 hours for 120 days (n=10), and a control group that will receive placebo with the same organoleptic characteristics for the same period of time (n=10).

Participants:

20 Mexican patients with obesity from the metropolitan area of Guadalajara diagnosed according to WHO criteria (BMI between ≥30 and <40 kg/m2), both sexes, who agreed to participate in the protocol through informed consent, with no known co-mobilities, use of current medication or any contraindication.

Intervention:

Intervention group that received 1 capsule of 500 mg of Triticum aestivum every 12 hours for 120 days (n=10), and a control group that received placebo with the same organoleptic characteristics for the same period (n=10). Both groups received general lifestyle and dietary recommendations.

Outcome Measures:

Primary outcome measures included flow-mediated dilation and arterial stiffness assessed by wave pulse velocity using non-invasive techniques. Secondary outcome measures encompassed anthropometric and clinical parameters, as well as laboratory results, and molecular markers such as endothelin-1 and nitric oxide.

Data Collection:

Baseline and post-intervention data were collected through standardized assessments and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* Sex indistinct, age between 30 and 60 years, BMI ≥30 and <40 kg/m2, signed informed consent, eumenorrheic women with mechanical or definitive contraceptive method without hormonal treatment.

Exclusion Criteria:

* History of: liver disease, chronic kidney disease, thyroid disease, cancer, diagnosis of diabetes, hypertension, dyslipidemia, patients with antihypertensive and antidiabetic treatment, lipid-lowering drugs, dietary supplements, acute infectious processes, alcoholism and/or active smoking, current pregnancy or breastfeeding, history of drug intake, recent surgery (in the last 3 months), pacemaker implantation, or any other permanent bioelectronic or metallic element that may modify the bioimpedance reading or may be affected by it.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Wave Pulse Velocity | 12 weeks
  The transit time of an aortic pressure wave between the common carotid artery and the common femoral artery. It is a standard measure of arterial stiffness.
Flow-mediated dilatation | 12 weeks
  Ecosonographic assessment of diameter changes in of the brachial artery secondary to increased blood flow.

SECONDARY OUTCOMES:
Body Max Index | 12 weeks
  An indicator of body density as determined by the relationship of body weight to body height. BMI=weight (kg)/height squared (m2). BMI correlates with body fat (adipose tissue). Their relationship varies with age and gender. For adults, BMI falls into these categories: below 18.5 (underweight); 18.5-24.9 (normal); 25.0-29.9 (overweight); 30.0 and above (obese).
Blood Pressure | 12 weeks
  The blood pressure in the arteries. It is commonly measured with a sphygmomanometer on the upper arm which represents the arterial pressure in the brachial artery.
Waist Hip Ratio | 12 weeks
  The waist circumference measurement divided by the hip circumference measurement. For both men and women, a waist-to-hip ratio (WHR) of 1.0 or higher is considered "at risk" for undesirable health consequences, such as heart disease and ailments associated with overweight. A healthy WHR is 0.90 or less for men, and 0.80 or less for women.
Medication Adherence | 12 weeks
  Voluntary cooperation of the patient in taking drugs or medicine as prescribed. This includes timing, dosage, and frequency.
Atherogenic Index | 12 weeks
  Logarithmically transformed ratio of molar concentrations of triglycerides to HDL-cholesterol

OTHER OUTCOMES:
Endotelin -1 Concentration | 12 weeks
  Plasma concentration of A 21-amino acid peptide produced in a variety of tissues including endothelial and vascular smooth-muscle cells, neurons and astrocytes in the central nervous system, and endometrial cells. It acts as a modulator of vasomotor tone, cell proliferation, and hormone production.
Nitric Oxide concentration | 12 weeks
  Plasma concentration of A free radical gas produced endogenously by a variety of mammalian cells, synthesized from arginine by nitric oxide synthase. Nitric oxide is one of the endothelium-dependent relaxing factors released by the vascular endothelium and mediates vasodilation. It also inhibits platelet aggregation, induces disaggregation of aggregated platelets, and inhibits platelet adhesion to the vascular endothelium. Nitric oxide activates cytosolic guanylate cyclase and thus elevates intracellular levels of cyclic GMP.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra O Hernández González, PhD, Principal Investigator — Instituto Mexicano del Seguro Social, Unidad de Investigación Biomédica 02.
Locations (1):
- Biomedical Unit Research 02, Specialties Hospital, Medical Unit of High Speciality, West National Medical Center, Mexican Social Security Institute., Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from the clinical investigation, except the personal identification of the subjects (name, address, teelephone, etc.)
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication.
Access Criteria: The data can be shared through a request addressed to the principal investigator Dr. Sandra Ofelia Hernández González, basing the reason for what they are requested.

REFERENCES:
- [Background] Kopustinskiene DM, Jakstas V, Savickas A, Bernatoniene J. Flavonoids as Anticancer Agents. Nutrients. 2020 Feb 12;12(2):457. doi: 10.3390/nu12020457. PMID 32059369
- [Background] Hostetler GL, Ralston RA, Schwartz SJ. Flavones: Food Sources, Bioavailability, Metabolism, and Bioactivity. Adv Nutr. 2017 May 15;8(3):423-435. doi: 10.3945/an.116.012948. Print 2017 May. PMID 28507008
- [Background] Bitew M, Desalegn T, Demissie TB, Belayneh A, Endale M, Eswaramoorthy R. Pharmacokinetics and drug-likeness of antidiabetic flavonoids: Molecular docking and DFT study. PLoS One. 2021 Dec 10;16(12):e0260853. doi: 10.1371/journal.pone.0260853. eCollection 2021. PMID 34890431
- [Background] Ciumarnean L, Milaciu MV, Runcan O, Vesa SC, Rachisan AL, Negrean V, Perne MG, Donca VI, Alexescu TG, Para I, Dogaru G. The Effects of Flavonoids in Cardiovascular Diseases. Molecules. 2020 Sep 21;25(18):4320. doi: 10.3390/molecules25184320. PMID 32967119
- [Background] Yamagata K, Yamori Y. Inhibition of Endothelial Dysfunction by Dietary Flavonoids and Preventive Effects Against Cardiovascular Disease. J Cardiovasc Pharmacol. 2020 Jan;75(1):1-9. doi: 10.1097/FJC.0000000000000757. PMID 31613843
- [Background] Rees A, Dodd GF, Spencer JPE. The Effects of Flavonoids on Cardiovascular Health: A Review of Human Intervention Trials and Implications for Cerebrovascular Function. Nutrients. 2018 Dec 1;10(12):1852. doi: 10.3390/nu10121852. PMID 30513729
- [Background] Micek A, Godos J, Del Rio D, Galvano F, Grosso G. Dietary Flavonoids and Cardiovascular Disease: A Comprehensive Dose-Response Meta-Analysis. Mol Nutr Food Res. 2021 Mar;65(6):e2001019. doi: 10.1002/mnfr.202001019. Epub 2021 Feb 25. PMID 33559970
- [Background] Yahfoufi N, Alsadi N, Jambi M, Matar C. The Immunomodulatory and Anti-Inflammatory Role of Polyphenols. Nutrients. 2018 Nov 2;10(11):1618. doi: 10.3390/nu10111618. PMID 30400131
- [Background] Luyen BT, Thao NP, Tai BH, Lim JY, Ki HH, Kim DK, Lee YM, Kim YH. Chemical constituents of Triticum aestivum and their effects on adipogenic differentiation of 3T3-L1 preadipocytes. Arch Pharm Res. 2015 Jun;38(6):1011-8. doi: 10.1007/s12272-014-0478-2. Epub 2014 Sep 23. PMID 25241774
- [Background] Poudel B, Nepali S, Xin M, Ki HH, Kim YH, Kim DK, Lee YM. Flavonoids from Triticum aestivum inhibit adipogenesis in 3T3-L1 cells by upregulating the insig pathway. Mol Med Rep. 2015 Aug;12(2):3139-45. doi: 10.3892/mmr.2015.3700. Epub 2015 Apr 29. PMID 25936595
- [Background] Im JY, Ki HH, Xin M, Kwon SU, Kim YH, Kim DK, Hong SP, Jin JS, Lee YM. Anti-obesity effect of Triticum aestivum sprout extract in high-fat-diet-induced obese mice. Biosci Biotechnol Biochem. 2015;79(7):1133-40. doi: 10.1080/09168451.2015.1006567. Epub 2015 Apr 30. PMID 25925980
- [Background] Bueno PCDS, Barbalho SM, Guiguer EL, Souza MDSS, Medeiros IRA, Zattiti IV, Bueno MDS, Nutels GS, Goulart RA, Araujo AC. Effects of Green Wheat (Triticum turgidum) and Common Wheat (Triticum aestivum) on the Metabolic Profile of Wistar Rats. J Med Food. 2019 Dec;22(12):1222-1225. doi: 10.1089/jmf.2019.0089. Epub 2019 Jul 18. PMID 31329009
- [Background] Naranjo CA, Busto U, Sellers EM, Sandor P, Ruiz I, Roberts EA, Janecek E, Domecq C, Greenblatt DJ. A method for estimating the probability of adverse drug reactions. Clin Pharmacol Ther. 1981 Aug;30(2):239-45. doi: 10.1038/clpt.1981.154. No abstract available. PMID 7249508
- [Background] Townsend RR. Arterial Stiffness: Recommendations and Standardization. Pulse (Basel). 2017 Jan;4(Suppl 1):3-7. doi: 10.1159/000448454. Epub 2016 Dec 23. PMID 28275588
- [Background] Daiber A, Steven S, Weber A, Shuvaev VV, Muzykantov VR, Laher I, Li H, Lamas S, Munzel T. Targeting vascular (endothelial) dysfunction. Br J Pharmacol. 2017 Jun;174(12):1591-1619. doi: 10.1111/bph.13517. Epub 2016 Jul 4. PMID 27187006
- [Background] Aroor AR, Jia G, Sowers JR. Cellular mechanisms underlying obesity-induced arterial stiffness. Am J Physiol Regul Integr Comp Physiol. 2018 Mar 1;314(3):R387-R398. doi: 10.1152/ajpregu.00235.2016. Epub 2017 Nov 22. PMID 29167167
- [Background] Para I, Albu A, Porojan MD. Adipokines and Arterial Stiffness in Obesity. Medicina (Kaunas). 2021 Jun 25;57(7):653. doi: 10.3390/medicina57070653. PMID 34202323
- [Background] Safar ME, Czernichow S, Blacher J. Obesity, arterial stiffness, and cardiovascular risk. J Am Soc Nephrol. 2006 Apr;17(4 Suppl 2):S109-11. doi: 10.1681/ASN.2005121321. PMID 16565231
- [Background] Zieman SJ, Melenovsky V, Kass DA. Mechanisms, pathophysiology, and therapy of arterial stiffness. Arterioscler Thromb Vasc Biol. 2005 May;25(5):932-43. doi: 10.1161/01.ATV.0000160548.78317.29. Epub 2005 Feb 24. PMID 15731494
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Thanassoulis G, Massaro JM, Corsini E, Rogers I, Schlett CL, Meigs JB, Hoffmann U, O'Donnell CJ, Fox CS. Periaortic adipose tissue and aortic dimensions in the Framingham Heart Study. J Am Heart Assoc. 2012 Dec;1(6):e000885. doi: 10.1161/JAHA.112.000885. Epub 2012 Dec 19. PMID 23316310
- [Background] Koenen M, Hill MA, Cohen P, Sowers JR. Obesity, Adipose Tissue and Vascular Dysfunction. Circ Res. 2021 Apr 2;128(7):951-968. doi: 10.1161/CIRCRESAHA.121.318093. Epub 2021 Apr 1. PMID 33793327
- [Background] Khan SS, Ning H, Wilkins JT, Allen N, Carnethon M, Berry JD, Sweis RN, Lloyd-Jones DM. Association of Body Mass Index With Lifetime Risk of Cardiovascular Disease and Compression of Morbidity. JAMA Cardiol. 2018 Apr 1;3(4):280-287. doi: 10.1001/jamacardio.2018.0022. PMID 29490333
- [Background] Powell-Wiley TM, Poirier P, Burke LE, Despres JP, Gordon-Larsen P, Lavie CJ, Lear SA, Ndumele CE, Neeland IJ, Sanders P, St-Onge MP; American Heart Association Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology; Council on Epidemiology and Prevention; and Stroke Council. Obesity and Cardiovascular Disease: A Scientific Statement From the American Heart Association. Circulation. 2021 May 25;143(21):e984-e1010. doi: 10.1161/CIR.0000000000000973. Epub 2021 Apr 22. PMID 33882682
- [Background] Lin X, Li H. Obesity: Epidemiology, Pathophysiology, and Therapeutics. Front Endocrinol (Lausanne). 2021 Sep 6;12:706978. doi: 10.3389/fendo.2021.706978. eCollection 2021. PMID 34552557
- See also: Cardiovascular Diseases — https://www.who.int/health-topics/cardiovascular-diseases
- See also: What Is Cardiovascular Disease. — https://world-heart-federation.org/what-is-cvd/
- See also: Atención oportuna, fundamental para prevenir y atender enfermedades cardiovasculares. — https://www.gob.mx/salud/es/articulos/atencion-oportuna-fundamental-para-prevenir-y-atender-enfermedades-cardiovasculares?idiom=es
- See also: Obesity and Overweight. — http://www.cenaprece.salud.gob.mx/descargas/pdf/PAE_PrevencionControlObesidadRiesgoCardiovascular2013_2018.pdf
- See also: Programa de Acción Específico Prevención y Control de la Obesidad y Riesgo Cardiovascular 2013-2018 — http://www.cenaprece.salud.gob.mx/descargas/pdf/PAE_PrevencionControlObesidadRiesgoCardiovascular2013_2018.pdf
- See also: Sobrepeso y Obesidad: factores de riesgo para desarrollar diabetes. México. — https://www.gob.mx/salud/articulos/sobrepeso-y-obesidad-factores-de-riesgos-para-desarrollar-diabetes